CLINICAL TRIAL: NCT02597309
Title: The Effect of add-on Canagliflozin in Patients With Type 2 Diabetes Treated With ≥200 Units Per Day of U-500 Insulin
Brief Title: The Effect of add-on Canagliflozin in Patients With Type 2 Diabetes Treated With U-500 Insulin
Acronym: I-Can
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Principal Investigator, Osama Hamdy, Medical Director, Obesity Clinical Program, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHS# 2015-03
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Diabetes, Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Intervention Group (Active Comparator): Subjects in this group will take canagliflozin in addition to their regular U-500 insulin dose and other antihyperglycemic medications. Canagliflozin dose will be titrated after 2 weeks from 100 mg once daily to 300 mg once daily. This dose will continue for 22 weeks.
  Interventions: Drug: Canagliflozin
- Control Group (Placebo Comparator): Subjects in this group will take a matched placebo in addition to their regular U-500 insulin dose and other antihyperglycemic medications for 2 weeks then another matched-placebo for 22 weeks.
  Interventions: Drug: Canagliflozin

INTERVENTIONS:
Drug: Canagliflozin
  Other Names: Invokana

SUMMARY:
The aim of this study is to evaluate the effect of adding a SGLT-2 inhibitor (namely Canagliflozin) on the dose of U-500 insulin required to achieve glycemic control in patients with type 2 diabetes. We hypothesize that adding Canagliflozin to patients treated with U-500 insulin may result in significant reduction in insulin dose due to improved insulin sensitivity and weight loss.

DETAILED DESCRIPTION:
Insulin resistance is one of the main causes of type 2 diabetes. Continuation of insulin resistance may lead to the failure of multiple oral antihyperglycemic medications in achieving glycemic control and the further requirement of escalading doses of insulin. On contrary, reduction of glucose toxicity and weight loss improves insulin sensitivity and may result in substantial reduction in insulin dose and %A1C.

U-500 insulin is the fastest-growing prescribed insulin in the US due to increased prevalence of severe obesity and extreme insulin resistance. Patients requiring high insulin doses of ≥200 units/day are the typical candidates for U-500 insulin. However, patients on such high doses of insulin rarely achieve target glycemic control.

Sodium-glucose co-transporter-2 (SGLT2) inhibitors are new antihyperglycemic medications approved for treatment of type 2 diabetes. Adding a SGLT-2 inhibitors to other antihyperglycemic medications was shown to reduce glucose toxicity, improve insulin sensitivity and reduce body weight. Consequently, daily insulin dose may be reduced without compromising glycemic control.

Canagliflozin is a sodium-glucose transporter subtype 2 (SGLT2) inhibitor that was approved by the FDA for the treatment of Type 2 diabetes in March, 2013. Canagliflozin, at the doses of 100mg and 300mg daily, improves blood sugar control by a novel mechanism which causes the kidneys to block reabsorption of about 50-80 grams of glucose. Canagliflozin lowers the renal threshold for glycosuria and causes excess glucose to be excreted in the urine.

The aim of this study is to evaluate the effect of adding a SGLT-2 inhibitor (namely Canagliflozin) on the dose of U-500 insulin required to achieve glycemic control in patients with type 2 diabetes. We hypothesize that adding Canagliflozin to patients treated with U-500 insulin may result in significant reduction in insulin dose due to improved insulin sensitivity and weight loss.

This is a double-blind, randomized, placebo-controlled clinical trial. Eligible subjects are patients with type 2 diabetes treated with ≥200 units per day of U-500 insulin with or without other antihyperglycemic medications. Participants will be randomized in a 1:1 ratio to one of the following 2 study arms.

I. Intervention Group: Subjects in this group will take canagliflozin in addition to their regular U-500 insulin dose and other antihyperglycemic medications. Canagliflozin dose will be titrated after 2 weeks from 100 mg once daily to 300 mg once daily. This dose will continue for 22 weeks.

II. Control Group: Subjects in this group will take a matched placebo in addition to their regular U-500 insulin dose and other antihyperglycemic medications for 2 weeks then another matched-placebo for 22 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject with type 2 diabetes
* Subject is managed on ≥200 units of U-500 insulin plus or minus stable dose of oral antihyperglycemic medications for at least 3 months (dose of oral antihyperglycemic medications will remain stable during intervention)
* Subject is male or non-pregnant and non-lactating female
* Subject with BMI > 25 kg/m2
* Subject with A1C >7%
* Subject with serum potassium between 5-5.5 mEq/L
* If subject is on chronic medications such as anti-hypertensive, lipid-lowering medications, thyroid medication or hormonal therapy, the dose of these medications should be stable for at least three months prior to the screening visit. These medications will not be changed during the intervention period unless mandatory

Exclusion Criteria:

* Subject has history of renal disease (serum creatinine >1.5mg/dL or GFR <60 mL/min/1.73 m2).
* Subject has history of recurrent urinary tract infections
* Subject has history of urinary incontinence
* Subject has history of prostate hypertrophy
* Subject has history of cancer bladder or cancer prostate
* Subject has history of hematuria
* Subject using corticosteroid treatment, except inhaled or topical steroids
* Subject having an active malignancy (excluding the following dermal malignancies: basal cell carcinoma, squamous cell carcinoma, carcinoma in-situ of the cervix).
* Subject states that he/she had a recent cardiovascular event (e.g. myocardial infarction, stroke) ≤ six months prior to the screening visit; or stated that he/she had history of congestive heart failure.
* Subject has hepatic failure or had status post organ transplant
* Subject has any chronic, contagious or infectious diseases
* Subject has blood clotting or bleeding disorders

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Reduction in insulin recuirement | Twenty four weeks
  Reduction in insulin requirements after adding canagliflozin with a difference in insulin dose of ≥30% between the 2 intervention groups

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States